CLINICAL TRIAL: NCT06636942
Title: Effects of Intermittent Pneumatic Compression Following an Officiall Soccer Match on Elite Youth Soccer Players
Brief Title: Effects of Intermittent Pneumatic Compression Following an Officiall Soccer Match
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maia (Other)
Responsible Party: Principal Investigator, Filipe Silvano Pinto Maia, Principal investigator, University of Maia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PDFM_004
Record Dates: First submitted 2024-10-02; First posted 2024-10-15 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Intermittent Pneumatic Compression; Placebo - Control
Keywords: sports; recovery; athletic performance; soccer
MeSH Terms: interventions — Intermittent Pneumatic Compression Devices

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intermittent pneumatic compression (Experimental): 30 minutes of intermittent pneumatic compression at 200mmHg
  Interventions: Device: Intermittent pneumatic compression
- Placebo (Placebo Comparator): A hydrant cream on a pad will be placed on participants quadriceps stating that they are using an inovative recovery cream.
  Interventions: Device: Intermittent pneumatic compression

INTERVENTIONS:
Device: Intermittent pneumatic compression — Following a soccer match, athletes will be enrolled in a recovery treatment: placebo intervention or intermittent pneumatic compression. Participants will be randomly assigned to each group. Neuromuscular tests (cmj) and perceptual questionnaires (hooper index) will be conducted.

SUMMARY:
This study aims to identify the effects of the use of intermittent pneumatic compression on the recovery kinetics following an official soccer match, in comparision with a placebo condition. Participants will perform neuromuscular tests (ie, cmj, low-frequency fatigue), respond to perception scales (RPE, perceived fatigue, soreness, sleep), and biochemical tests (CK analysis). These assessments will be carried out before the match, 30 minutes post match, at the 24th and 48th hour.

ELIGIBILITY:
Inclusion Criteria:

* elite soccer players

Exclusion Criteria:

* absent from injuries
* playing less than 70 minutes

Ages: 18 Years to 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-06-29 (Actual)

PRIMARY OUTCOMES:
Countermovement jump height | 30 minute, 24 hour, 48 hour
  Height measure using CMJ test
low-frequency fatigue | baseline, 30 minute, 24 hour, and 48 hour
  LFF measured using Myocene (Liege, Belgium)
creatine-kinase | baseline, 24 hour, and 48 hour
  Muscle damage asses using the biomarker CK
Hooper index | baseline, 30 minute, 24 hour, and 48 hour
  Application of the hooper index questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade da Maia, Maia, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Maia F, Tito S, Correia M, Nakamura FY, Ribeiro J. Intermittent pneumatic compression does not improve post-match neuromuscular, biochemical or perceptual recovery in international-level youth soccer players: a randomized placebo-controlled trial. BMC Sports Sci Med Rehabil. 2026 Feb 9. doi: 10.1186/s13102-026-01580-5. Online ahead of print. PMID 41656279